CLINICAL TRIAL: NCT02596490
Title: Couple-Based Meditation for Metastatic Lung Cancer Patients and Their Partners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0275; 1R21CA191711 (NIH); NCI-2015-02128 (Registry Identifier: NCI CTRP-Clinical Trials Registry)
Record Dates: First submitted 2015-10-29; First posted 2015-11-04 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Couples-based meditation program; Couples-based cancer-related discussion program; Questionnaires; Surveys; Metastatic lung cancer; Quality of life; QOL
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Surveys and Questionnaires; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1: Couple-Based Mindfulness Disclosure Group (Experimental): Phase 1:
  Couples participate in 2 guided meditation sessions. During the sessions, participants do deep breathing and visualization exercises then asked to review the exercises. Participants also asked for feedback about the instructions. Participants complete a written review about the program and a questionnaire about their general health and well-being. Each session will last about 60-90 minutes.
  Interventions: Behavioral: Questionnaires; Behavioral: Meditation and Discussion Sessions
- Phase 2: Couple-Based Mindfulness Disclosure Group (Experimental): Phase 2:
  Participants complete 12 questionnaires before first meditation and discussion session. Questionnaires ask about participant's health, mood, level of fatigue, sleeping habits, relationship, and their quality of life. It should take about 45 minutes to complete these questionnaires. After completing the last session, about 4 weeks later, participants complete the same questionnaires again. Participants also complete a program review.
  Couples participate in 4 guided meditation sessions with a trained meditation instructor. Participants do deep breathing and visualization exercises. All meditation and discussion sessions videotaped.
  Participants continue daily meditation practice and some other short exercises at home.
  Interventions: Behavioral: Questionnaires; Behavioral: Meditation and Discussion Sessions
- Phase 3: Couple-Based Mindfulness Disclosure Group (Experimental): Participant completes 13 questionnaires before first mediation session, after last session, and again 3 months later. Questionnaires ask about participant's health, any symptoms they may be having, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. Partners complete 12 questionnaires about their health, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. It should take about 45 minutes to complete these questionnaires.
  Participant and partner attend meditation class with a trained meditation instructor each week for 4 weeks. Each session will last about 60 minutes total. Meditation and discussion sessions videotaped.
  Interventions: Behavioral: Questionnaires; Behavioral: Meditation and Discussion Sessions
- Phase 3: Cancer-Related Discussion Program Group (Experimental): Participant completes 13 questionnaires before first mediation session, after last session, and again 3 months later. Questionnaires ask about participant's health, any symptoms they may be having, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. Partners complete 12 questionnaires about their health, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. It should take about 45 minutes to complete these questionnaires.
  Participant and partner take part in a discussion program, 1 discussion session each week for 4 weeks with a trained interventionist. These are one-on-one sessions. Issues discussed for couples coping with cancer. Each session will last about 60 minutes.
  Interventions: Behavioral: Questionnaires; Behavioral: Cancer-Related Discussion Program
- Phase 3: Attention Control (AC) Group (Other): Participant completes 13 questionnaires at baseline and again 3 months later. Questionnaires ask about participant's health, any symptoms they may be having, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. Partners complete 12 questionnaires about their health, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. It should take about 45 minutes to complete these questionnaires.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Phase 1: At end of second meditation and discussion session, couples complete complete a written review about the program in general and a questionnaire about their general health and well-being.
  Phase 2: Couples complete 12 questionnaires before first meditation and discussion session. Questionnaires ask about participant's health, mood, level of fatigue, sleeping habits, their relationship, and quality of life. Same questionnaires completed 1 week after mediation sessions.
  Phase 3: Participant complete 13 questionnaires before first mediation session, after last session, and again 3 months later. Questionnaires ask about participant's health, any symptoms they may be having, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. Partners complete 12 questionnaires about their health, mood, level of fatigue, sleeping habits, their relationship, and their quality of life. AC group completes same questionnaires with no intervention.
  Other Names: Surveys
Behavioral: Meditation and Discussion Sessions — Phase 1: Participant and partner attend 2 meditation sessions with a mediation trained instructor. Each session will last about 60-90 minutes.
  Phase 2 and 3: Participant and partner attend meditation class with a trained meditation instructor each week for 4 weeks. Each session will last about 60 minutes total. Meditation and discussion sessions videotaped.
  Arms: Phase 1: Couple-Based Mindfulness Disclosure Group; Phase 2: Couple-Based Mindfulness Disclosure Group; Phase 3: Couple-Based Mindfulness Disclosure Group
Behavioral: Cancer-Related Discussion Program — Phase 3: Participant and partner attend 1 discussion session each week for 4 weeks with a trained interventionist. During the discussion sessions, participants discuss issues for couples coping with cancer. Each session will last about 60 minutes.
  Arms: Phase 3: Cancer-Related Discussion Program Group

SUMMARY:
Objectives:

Our specific aims are to:

Aim 1: Examine the feasibility of a couple-based meditation program in 50 patients with metastatic lung cancer and their partners.

Aim 2: Establish the initial efficacy of a couple-based meditation program in patients and their partners regarding physical, psychological, and spiritual quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. ALL PHASES, PATIENTS ONLY: Diagnosed with stage IV Non-Small Cell Lung Cancer (NSCLC)
2. ALL PHASES, PATIENTS ONLY: Currently receiving treatment (e.g. radiotherapy, chemotherapy) at MD Anderson Cancer Center
3. ALL PHASES, PATIENTS ONLY: Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
4. ALL PHASES, PATIENTS ONLY: Have a romantic partner with whom they have resided for a minimum of 6 months
5. ALL PHASES, PATIENTS AND PARTNERS: Must be at least 18 years old
6. ALL PHASES, PATIENTS AND PARTNERS: Able to read and speak English
7. ALL PHASES, PATIENTS AND PARTNERS: Able to provide consent.

Exclusion Criteria:

1. ALL PHASES, PATIENTS AND PARTNERS: Not oriented to time, place, or person as deemed by the clinical team
2. ALL PHASES, PATIENTS AND PARTNERS: Regular (self-defined) participation in psychotherapy or a formal cancer support group
3. ALL PHASES, PATIENTS AND PARTNERS: Prior enrollment in a couple-based mind-body intervention research study (protocols 2011-1179, 2013-0496, 2014-0036) conducted by the principal investigator including phase 1 or phase 2 of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-04-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Couple-Based Meditation for Participants with Lung Cancer and Their Partners | 4 months
  Efficacy based on physical, psychological, and spiritual quality of life outcomes.
  T-tests used to compare the pre-post change in the quality of life (QOL) outcomes between interventions separately for the participants and caregivers.
Feasibility of Couple-Based Meditation for Participants with Lung Cancer and Their Partners | 4 months
  Intervention deemed feasible if >60% of enrolled couples complete Time 1 and Time 2 survey assessments.
Feasibility of Couple-Based Meditation for Participants with Lung Cancer and Their Partners | 4 months
  Intervention deemed feasible if on average >50% of all practice sessions are attended.
Feasibility of Couple-Based Meditation for Participants with Lung Cancer and Their Partners | 4 months
  Intervention deemed feasible if no attributable adverse events (AE) or serious adverse events (SAE) occur.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, PHD, MA, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Memorial Hermann, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Milbury K, Tsao AS, Liao Z, Owns A, Engle R, Gonzalez EA, Bruera E, Cohen L. A research protocol for a pilot randomized controlled trial designed to examine the feasibility of a couple-based mind-body intervention for patients with metastatic lung cancer and their partners. Pilot Feasibility Stud. 2018 Jan 24;4:37. doi: 10.1186/s40814-018-0231-6. eCollection 2018. PMID 29416870
- See also: MD Anderson Cancer Center — http://www.mdanderson.org